CLINICAL TRIAL: NCT07137728
Title: A Randomized Controlled Trial to Evaluate the Effect of Dual Frequency Low-Level Laser Therapy on Pain Intensity, Pressure Pain Threshold, and Functional Outcomes in Patients With Myofascial Trigger Points in the Upper Trapezius Muscle
Brief Title: Dual Frequency Low-Level Laser Therapy in Myofascial Trigger Points of Upper Trapezius
Acronym: DF-LLLT-MTP-UT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0006
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Myofascial Pain Syndrome (MPS); Upper Trapezius Muscle Pain
Keywords: Low-Level Lazer Therapy; Dual Frequency Laser; Upper Trapezius Muscle; Myofascial Trigger Points; Myofascial Pain Syndrome; Neck Pain; Photobiomodulation; Physical Therapy Intervention
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two groups:
  1. Experimental group:
     Dual frequency low-level laser therapy plus conventional therapy.
  2. Control group:
  Sham laser therapy plus conventional therapy.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation. The sham laser device will look and sound identical to the active device but will not emit therapeutic light, ensuring participants are unaware of their group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Frequency Low-Level Laser Therapy + Conventional Therapy (Experimental): Participants will receive dual frequency low-level laser therapy (DF-LLLT) at 830 nm, 100 mW/cm², 9.12 Hz, 5 J/cm², applied perpendicularly over each identified myofascial trigger point in the upper trapezius muscle for 3 minutes 9 seconds per point, twice weekly for 4 weeks. In addition, they will perform a standardized stretching and strengthening exercise program for the neck and shoulders.
  Interventions: Device: Dual Frequency Low-Level Laser Therapy; Other: Conventional Therapy (Stretching and Strengthening Program)
- Sham Laser + Conventional Therapy (Placebo Comparator): Participants will receive sham laser therapy with identical appearance, sounds, and application time as the experimental laser but without light emission. In addition, they will perform the same standardized stretching and strengthening exercise program for the neck and shoulders.
  Interventions: Device: Sham Laser; Other: Conventional Therapy (Stretching and Strengthening Program)

INTERVENTIONS:
Device: Dual Frequency Low-Level Laser Therapy — DF-LLLT (830 nm, 100 mW/cm², 9.12 Hz, 5 J/cm²) applied over each identified trigger point for 3 minutes 9 seconds per point, twice weekly for 4 weeks.
  Arms: Dual Frequency Low-Level Laser Therapy + Conventional Therapy
Device: Sham Laser — Inactive laser device identical in appearance and sound to the active laser but without light emission, applied for 3 minutes 9 seconds per point, twice weekly for 4 weeks.
  Arms: Sham Laser + Conventional Therapy
Other: Conventional Therapy (Stretching and Strengthening Program) — A standardized physiotherapy program including stretching and strengthening exercises for the cervical and shoulder muscles. The program is performed under physiotherapist supervision twice weekly for 4 weeks. Exercises are identical across both study arms and include stretching of the upper trapezius and strengthening of the neck and scapular stabilizer muscles.

SUMMARY:
The goal of this clinical trial is to learn if dual frequency low-level laser therapy (DF-LLLT) works to reduce pain and improve neck function in adults with myofascial trigger points in the upper trapezius muscle. It will also determine whether DF-LLLT improves cervical range of motion.

The main questions it aims to answer are:

i)Does DF-LLLT reduce pain intensity on the Visual Analog Scale (VAS) more than sham laser therapy? ii)Does DF-LLLT improve functional status (Neck Disability Index) and cervical range of motion more than sham laser therapy?

Researchers will compare DF-LLLT plus conventional therapy to sham laser plus conventional therapy to see if DF-LLLT has greater therapeutic effects.

Participants will:

1. Receive either DF-LLLT or sham laser therapy twice weekly for 4 weeks
2. Perform a standardized stretching and strengthening exercise program for the neck and shoulders.
3. Attend clinic visits at baseline, week 2, and week 4 for assessments of pain, function, and cervical mobility.

DETAILED DESCRIPTION:
Myofascial trigger points (MTrPs) in the upper trapezius muscle are a frequent source of neck pain, muscle stiffness, and reduced cervical mobility. They are characterized by hypersensitive palpable nodules within taut muscle fibers that can produce local and referred pain. Traditional management strategies include stretching, strengthening, and various physical therapy modalities, but recurrence and incomplete relief are common.

Low-level laser therapy (LLLT) is a non-invasive photobiomodulation technique shown to reduce pain and inflammation and promote tissue healing. Dual frequency LLLT may provide enhanced therapeutic effects compared to single frequency LLLT by delivering both continuous and pulsed light energy to targeted tissues. However, clinical evidence for its use in upper trapezius MTrPs is limited.

This single-blinded randomized controlled trial will recruit 32 male and female participants aged 20-55 years who meet the diagnostic criteria for MTrPs according to Simons' guidelines. Participants will be randomly assigned to one of two groups:

Experimental group: DF-LLLT (830 nm, 100 mW/cm², 9.12 Hz, 5 J/cm²) applied perpendicularly over each identified MTrP for 3 minutes 9 seconds per point, twice weekly for 4 weeks, plus a standardized stretching and strengthening program.

Control group: Sham laser therapy with identical appearance and application time but without light emission, plus the same exercise program.

Primary and secondary outcomes will be assessed at baseline, week 2, and week 4:

Primary outcome: Change in pain intensity measured using the Visual Analog Scale (VAS)

Secondary outcomes: Change in functional status (Neck Disability Index) and change in cervical range of motion (flexion, extension, lateral flexion, and rotation) measured with a goniometer.

The study aims to determine whether DF-LLLT provides superior pain relief, functional improvement, and mobility gains compared to sham laser therapy when combined with conventional exercises. Statistical analysis will be performed using SPSS 21.0, with significance set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria: This includes the following;

* Men and women aged 20-55 years.
* Diagnosis of myofascial pain based on Simons criteria.
* At least two trigger points in the upper trapezius muscle.
* Pain duration ≥ 3 months.
* VAS pain score ≥ 5.
* Limited cervical range of motion due to trigger points.

Exclusion Criteria: The exclusion Criteria is given below;

* Pregnancy.
* Use of anticoagulants.
* Bleeding disorders or dermatological diseases at treatment site.
* History of infectious, inflammatory, tumoral, cardiopulmonary, psychiatric, or systemic diseases.
* Kellgren stage 3-4 cervical osteoarthritis or cervical disc herniation causing radiculopathy.
* Diagnosis of fibromyalgia.
* Inability to follow instructions or complete questionnaires.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale) | Baseline, Week 2, Week 4
  Change in pain intensity as measured by a 10 cm Visual Analog Scale (0 = no pain, 10 = worst imaginable pain).

SECONDARY OUTCOMES:
Functional Status (Neck Disability Index) | Baseline, Week 2, Week 4
  Change in functional disability as measured by the Neck Disability Index, a validated questionnaire scored from 0 to 50, where higher scores indicate greater disability.
Cervical Range of Motion (CROM) | Baseline, Week 2, Week 4
  Change in cervical range of motion including flexion, extension, right and left lateral flexion, and right and left rotation, measured with a universal goniometer.